CLINICAL TRIAL: NCT05437874
Title: Effects of Carbonated Beverage Consumption on Oral pH and Bacterial Proliferation in Adolescents: A Randomized Crossover Clinical Trial.
Brief Title: Carbonated Beverage Consumption in pH and Bacterial Proliferation
Acronym: pHSB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Guadalupe Barajas, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HIM 2017-084 SSA 1411
Record Dates: First submitted 2022-06-09; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: pH; Saliva; Dental Plaque
Keywords: pH; caries; saliva; artificial sweetener; carbonated beverages; dental biofilm
MeSH Terms: conditions — Dental Plaque | interventions — Natural Childbirth

STUDY DESIGN:
Intervention Model Description: A Randomized Crossover Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: colors were designated for each drink
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Natural Water (Placebo Comparator): 355 ml of water should be drunk.
  * Salivary pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Dental biofilm pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Streptococcus mutans dental biofilm formation ( Colony Forming Units) will be conducted at 0 and 120 minutes later
  Interventions: Drug: Natural Water
- Carbonated water (Active Comparator): 355 ml of carbonated water should be drunk
  * Salivary pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Dental biofilm pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Streptococcus mutans dental biofilm formation ( Colony Forming Units) will be conducted at 0 and 120 minutes later
  Interventions: Drug: Natural Water
- Aspartame/acesulfame K (Experimental): 355 ml of drink of diet coke should be drunk.
  * Salivary pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Dental biofilm pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Streptococcus mutans dental biofilm formation ( Colony Forming Units) will be conducted at 0 and 120 minutes later
  Interventions: Drug: Natural Water
- Saccharose (Experimental): 355 ml of drink of regular coke should be drunk
  * Salivary pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Dental biofilm pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Streptococcus mutans dental biofilm formation ( Colony Forming Units) will be conducted at 0 and 120 minutes later
  Interventions: Drug: Natural Water

INTERVENTIONS:
Drug: Natural Water — 355 ml of regular coke, diet coke or mineral water should be drunk.
  * Salivary pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Dental biofilm pH will be determined at 0, 5, 10, 15, 30, 45 and 60 minutes later
  * Streptococcus mutans dental biofilm formation ( Colony Forming Units) will be conducted at 0 and 120 minutes later
  Other Names: Plain water

SUMMARY:
The objective of this research is to evaluate the oral modifications caused by different types of coke drinks (regular coke and diet coke). The salivary and the dental biofilm pH will be determined in the first minutes after their consumption. Additionally, the bacterial proliferation of dental biofilm will be evaluated.

DETAILED DESCRIPTION:
Sugary soft drinks modify oral pH and favor bacterial proliferation and are associated with the development of caries. Information on the effects of consuming carbonated drinks without sucrose is limited.

In this crossover clinical trial, salivary pH and dental biofilm pH will be determined. These will be registered at 0, 5, 10, 15, 30, 45, and 60 min after the participants ingested 355 ml of natural water, soft drink with sucrose, soft drink with aspartame/acesulfame K or carbonated water on different days (1 week between each other). In addition, dental biofilm cultures will be conducted at 0 and 120 minutes after intake of each beverage to determine Streptococcus mutans biofilm formation.

The patients will be invited to participate and informed of the potential risks. Those who signed informed consent and have eligibility requirements will be randomized in a double-blind manner.

The data collection will be carried out in records forms, including verifying the patient's previous conditions, identification data (ID, age, gender,) and possible adverse events. If any adverse effect could exist, the research team will be notified for the implementation of possible changes.

A HANNA HI 221 potentiometer (HANNA Instruments Inc. Woonsocket-RI-USA, Romania) will be used to determine salivary pH and dental biofilm pH. The electrode will be calibrated using buffer solutions of pH 4.0 and 7.0 for correct records. The electrode will be washed with distilled water before and after each sample. The data will be collected by 2 verifiers, guaranteeing that the information obtained is the same as that indicated on the potentiometer; a stopwatch will indicate the exact time for obtaining the pH values.

Samples of dental biofilm will be taken, and Streptococcus mutans biofilm formation will be evaluated at 0 and 120 minutes after taking each beverage. The samples will be cultivated in suitable conditions, identified and compared with ATCC. The samples obtained will be analyzed in the same place of collection to avoid possible contamination.

Sample size with an alpha=0.05 and a beta=0.8 include 22, considering 20% losses.

Variables will be described with frequencies and percentages or medians and interquartile range (IQR) according to the variable type. Salivary pH and dental biofilm at different times will be compared using ANOVA analysis with adjustment for multiple comparisons using Bonferroni correction. Changes in the bacterial proliferation of the dental biofilm at 0 and 120 min will be compared using the Wilcoxon test and intergroup changes will be compared using the Kruskal-Wallis test. The statistical program SPSS v. 22 will be used and statistical significance will be considered with a p ≤ 0.05

ELIGIBILITY:
Inclusion Criteria:

* Habitual consumption of soft drinks
* DMFT (Decayed, Missing, and Filled Teeth) index of at least 3
* Agree to participate in the study and sign informed consent
* Parents sign informed consent
* Any nutritional condition

Exclusion Criteria:

* Undergoing orthodontic treatment
* Received a topical application of fluoride during the last 3 months
* Having a motor disability that interfered with tooth brushing
* Consuming drugs or being carriers of diseases that cause xerostomia
* Being under antibiotic therapy during the study period
* Having active periodontal infections.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Mean salivary pH with regular coke | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with regular coke | 60 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with diet coke | 60 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with carbonated water | 60 minutes
  logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natual water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 60 minutes
  Logarithm of hydrogen ion concentration

SECONDARY OUTCOMES:
Mean dental biofilm pH with regular coke | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with regular coke | 60 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental pH biofilm with diet coke | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet coke | 60 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with carbonated water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with diet carbonated water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with carbonated water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with carbonated water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental pellicle pH with carbonated water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with carbonated water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with carbonated water | 60 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 60 minutes
  Logarithm of hydrogen ion concentration

OTHER OUTCOMES:
Mean Colony Forming Units Streptococcus mutans dental biofilm with regular coke | 0 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with regular coke | 120 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with diet coke | 0 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with diet coke | 120 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with carbonated water | 0 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with carbonated water | 120 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with natural water | 0 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.
Mean Colony Forming Units Streptococcus mutans dental biofilm with natural water | 120 minutes
  Number of viable colonies on a semisolid agar culture medium that are visible and separable.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Garduño, MSc., PhD, Study Director — Children´s Hospital of Mexico Federico Gómez
Locations (1):
- Children´s Hospital of Mexico Federico Gómez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: SAP
Time Frame: when summary data are published
Access Criteria: The data will be shared with researchers interested in data analysis, request to email: americaml@hotmail.com, review of the request by MSc., PhD. America Liliana Miranda Lora
URL: https://drive.google.com/drive/folders/1d_1HgpcKEtQPmhMwOtco58yui3CWh7j3?usp=sharing

REFERENCES:
- [Background] Gonzalez-Aragon Pineda AE, Garcia Perez A, Garcia-Godoy F. Salivary parameters and oral health status amongst adolescents in Mexico. BMC Oral Health. 2020 Jul 6;20(1):190. doi: 10.1186/s12903-020-01182-8. PMID 32631313
- [Background] Machiulskiene V, Campus G, Carvalho JC, Dige I, Ekstrand KR, Jablonski-Momeni A, Maltz M, Manton DJ, Martignon S, Martinez-Mier EA, Pitts NB, Schulte AG, Splieth CH, Tenuta LMA, Ferreira Zandona A, Nyvad B. Terminology of Dental Caries and Dental Caries Management: Consensus Report of a Workshop Organized by ORCA and Cariology Research Group of IADR. Caries Res. 2020;54(1):7-14. doi: 10.1159/000503309. Epub 2019 Oct 7. PMID 31590168
- [Background] Vieira AR, Modesto A, Marazita ML. Caries: review of human genetics research. Caries Res. 2014;48(5):491-506. doi: 10.1159/000358333. Epub 2014 May 21. PMID 24853115
- [Background] Krzysciak W, Pluskwa KK, Piatkowski J, Krzysciak P, Jurczak A, Koscielniak D, Skalniak A. The usefulness of biotyping in the determination of selected pathogenicity determinants in Streptococcus mutans. BMC Microbiol. 2014 Aug 5;14:194. doi: 10.1186/1471-2180-14-194. PMID 25096795
- [Background] Mathur MR, Tsakos G, Millett C, Arora M, Watt R. Socioeconomic inequalities in dental caries and their determinants in adolescents in New Delhi, India. BMJ Open. 2014 Dec 12;4(12):e006391. doi: 10.1136/bmjopen-2014-006391. PMID 25500618
- [Background] Koo H, Falsetta ML, Klein MI. The exopolysaccharide matrix: a virulence determinant of cariogenic biofilm. J Dent Res. 2013 Dec;92(12):1065-73. doi: 10.1177/0022034513504218. Epub 2013 Sep 17. PMID 24045647
- [Background] Gonzalez-Aragon Pineda AE, Borges-Yanez SA, Irigoyen-Camacho ME, Lussi A. Relationship between erosive tooth wear and beverage consumption among a group of schoolchildren in Mexico City. Clin Oral Investig. 2019 Feb;23(2):715-723. doi: 10.1007/s00784-018-2489-8. Epub 2018 May 13. PMID 29756172
- [Background] Lemos JA, Palmer SR, Zeng L, Wen ZT, Kajfasz JK, Freires IA, Abranches J, Brady LJ. The Biology of Streptococcus mutans. Microbiol Spectr. 2019 Jan;7(1):10.1128/microbiolspec.gpp3-0051-2018. doi: 10.1128/microbiolspec.GPP3-0051-2018. PMID 30657107
- [Background] Bechir F, Pacurar M, Tohati A, Bataga SM. Comparative Study of Salivary pH, Buffer Capacity, and Flow in Patients with and without Gastroesophageal Reflux Disease. Int J Environ Res Public Health. 2021 Dec 25;19(1):201. doi: 10.3390/ijerph19010201. PMID 35010461
- [Background] Peng X, Han Q, Zhou X, Chen Y, Huang X, Guo X, Peng R, Wang H, Peng X, Cheng L. Effect of pH-sensitive nanoparticles on inhibiting oral biofilms. Drug Deliv. 2022 Dec;29(1):561-573. doi: 10.1080/10717544.2022.2037788. PMID 35156501
- [Background] Foglio-Bonda PL, Brilli K, Pattarino F, Foglio-Bonda A. Salivary flow rate and pH in patients with oral pathologies. Eur Rev Med Pharmacol Sci. 2017 Jan;21(2):369-374. PMID 28165549
- [Background] Aiuchi H, Kitasako Y, Fukuda Y, Nakashima S, Burrow MF, Tagami J. Relationship between quantitative assessments of salivary buffering capacity and ion activity product for hydroxyapatite in relation to cariogenic potential. Aust Dent J. 2008 Jun;53(2):167-71. doi: 10.1111/j.1834-7819.2008.00027.x. PMID 18494973
- [Background] Ilie O, van Turnhout AG, van Loosdrecht MC, Picioreanu C. Numerical modelling of tooth enamel subsurface lesion formation induced by dental plaque. Caries Res. 2014;48(1):73-89. doi: 10.1159/000354123. Epub 2013 Nov 14. PMID 24248036
- [Background] Humphrey SP, Williamson RT. A review of saliva: normal composition, flow, and function. J Prosthet Dent. 2001 Feb;85(2):162-9. doi: 10.1067/mpr.2001.113778. PMID 11208206
- [Background] Kaur A, Kwatra KS, Kamboj P. Evaluation of non-microbial salivary caries activity parameters and salivary biochemical indicators in predicting dental caries. J Indian Soc Pedod Prev Dent. 2012 Jul-Sep;30(3):212-7. doi: 10.4103/0970-4388.105013. PMID 23263424
- [Background] Ahmadi-Motamayel F, Falsafi P, Goodarzi MT, Poorolajal J. Comparison of Salivary pH, Buffering Capacity and Alkaline Phosphatase in Smokers and Healthy Non-Smokers: Retrospective cohort study. Sultan Qaboos Univ Med J. 2016 Aug;16(3):e317-21. doi: 10.18295/squmj.2016.16.03.009. Epub 2016 Aug 19. PMID 27606111
- [Background] Gornowicz A, Tokajuk G, Bielawska A, Maciorkowska E, Jablonski R, Wojcicka A, Bielawski K. The assessment of sIgA, histatin-5, and lactoperoxidase levels in saliva of adolescents with dental caries. Med Sci Monit. 2014 Jun 29;20:1095-100. doi: 10.12659/MSM.890468. PMID 24974109
- [Background] Acquier AB, Pita AK, Busch L, Sanchez GA. Comparison of salivary levels of mucin and amylase and their relation with clinical parameters obtained from patients with aggressive and chronic periodontal disease. J Appl Oral Sci. 2015 May-Jun;23(3):288-94. doi: 10.1590/1678-775720140458. PMID 26221923
- [Background] Gabryel-Porowska H, Gornowicz A, Bielawska A, Wojcicka A, Maciorkowska E, Grabowska SZ, Bielawski K. Mucin levels in saliva of adolescents with dental caries. Med Sci Monit. 2014 Jan 18;20:72-7. doi: 10.12659/MSM.889718. PMID 24441930
- [Background] Hideaki W, Tatsuya H, Shogo M, Naruto Y, Hideaki T, Yoichi M, Yoshihiro O, Kazuo U, Hidenori T. Effect of 100 Hz electroacupuncture on salivary immunoglobulin A and the autonomic nervous system. Acupunct Med. 2015 Dec;33(6):451-6. doi: 10.1136/acupmed-2015-010784. Epub 2015 Oct 8. PMID 26449884
- [Background] Moradi G, Mohamadi Bolbanabad A, Moinafshar A, Adabi H, Sharafi M, Zareie B. Evaluation of Oral Health Status Based on the Decayed, Missing and Filled Teeth (DMFT) Index. Iran J Public Health. 2019 Nov;48(11):2050-2057. PMID 31970104
- [Result] Moynihan PJ, Kelly SA. Effect on caries of restricting sugars intake: systematic review to inform WHO guidelines. J Dent Res. 2014 Jan;93(1):8-18. doi: 10.1177/0022034513508954. Epub 2013 Dec 9. PMID 24323509
- [Result] Olivier B, Serge AH, Catherine A, Jacques B, Murielle B, Marie-Chantal CL, Sybil C, Jean-Philippe G, Sabine H, Esther K, Perrine N, Fabienne R, Gerard S, Irene M. Review of the nutritional benefits and risks related to intense sweeteners. Arch Public Health. 2015 Oct 1;73:41. doi: 10.1186/s13690-015-0092-x. eCollection 2015. PMID 26430511
- [Result] Brambilla E, Cagetti MG, Ionescu A, Campus G, Lingstrom P. An in vitro and in vivo comparison of the effect of Stevia rebaudiana extracts on different caries-related variables: a randomized controlled trial pilot study. Caries Res. 2014;48(1):19-23. doi: 10.1159/000351650. Epub 2013 Nov 6. PMID 24216624
- [Result] Jawale BA, Bendgude V, Mahuli AV, Dave B, Kulkarni H, Mittal S. Dental plaque pH variation with regular soft drink, diet soft drink and high energy drink: an in vivo study. J Contemp Dent Pract. 2012 Mar 1;13(2):201-4. doi: 10.5005/jp-journals-10024-1121. PMID 22665748
- [Result] Sanchez GA, Fernandez De Preliasco MV. Salivary pH changes during soft drinks consumption in children. Int J Paediatr Dent. 2003 Jul;13(4):251-7. doi: 10.1046/j.1365-263x.2003.00469.x. PMID 12834385
- [Result] Uma E, Theng KS, Yi LLH, Yun LH, Varghese E, Soe HHK. Comparison of Salivary pH Changes after Consumption of Two Sweetened Malaysian Local Drinks among Individuals with Low Caries Experience: A Pilot Study. Malays J Med Sci. 2018 Jul;25(4):100-111. doi: 10.21315/mjms2018.25.4.10. Epub 2018 Aug 30. PMID 30914852
- [Result] Roos EH, Donly KJ. In vivo dental plaque pH variation with regular and diet soft drinks. Pediatr Dent. 2002 Jul-Aug;24(4):350-3. PMID 12212881
- [Result] Llena-Puy C. The role of saliva in maintaining oral health and as an aid to diagnosis. Med Oral Patol Oral Cir Bucal. 2006 Aug;11(5):E449-55. English, Spanish. PMID 16878065
- [Result] Saeed S, Al-Tinawi M. Evaluation of acidity and total sugar content of children's popular beverages and their effect on plaque pH. J Indian Soc Pedod Prev Dent. 2010 Jul-Sep;28(3):189-92. doi: 10.4103/0970-4388.73783. PMID 21157052

DOCUMENTS (1):
  • Informed Consent Form (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT05437874/ICF_000.pdf